CLINICAL TRIAL: NCT04736797
Title: Transition in Transgender: Physiological Changes in Brain and Behavior
Brief Title: Transition in Transgender
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: RWTH Aachen University (Other)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Other Study IDs: 19-176
Record Dates: First submitted 2020-03-10; First posted 2021-02-03 (Actual); Last update posted 2021-02-12 (Actual); Status verified 2021-01

CONDITIONS: Gender Dysphoria
Keywords: Transgender; female to male; male to female; Hormone treatment; Gender reassignment
MeSH Terms: conditions — Gender Dysphoria

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: Transgender people who seek hormone treatment
- Control participants: volunteers without gender dysphoria

SUMMARY:
The aim of this longitudinal, observational study is to investigate the effects of gender-affirming hormone treatment in FTM (female to male) and MTF (male to female) transgender (TG) people with regard to changes in brain structure and function as well as psychological and behavioral consequences. Methodological problems and missing studies in this area were mentioned several times with an emphasis on the need for longitudinal research.

DETAILED DESCRIPTION:
Transgender (TG) is still a polarizing issue today. The lack of acceptance in society and often even in one's own family, the feeling of a lack of identity and connection with one's own body and the experienced discrimination all lead to a considerable degree of suffering in TG and elevated levels of psychiatric symptoms as well as a reduced quality of life. Many TG people seek hormonal treatment. Physical and psychological consequences of this treatment still need to be revealed.

To this aim, the investigators recruit TG people (MTF and FTM) who intend to seek gender-affirming hormonal treatment. Before treatment, various measures will be taken, including a semi-structured interview to assess psychiatric symptoms, self-ratings, behavioral experiments (to assess male/female face recognition and male/female voice perception), while functional MRI scans are taken to assess respective neural correlates. In addition, resting-state scans as well as anatomic images will be taken.

Six months after having started gender-affirming hormone treatment, participants will be reinvited to undergo the same study protocol.

In between testing sessions, patients will perform several online surveys regarding their psychological well-being.

ELIGIBILITY:
Inclusion Criteria:

1. a diagnosed gender dysphoria (DSM 5) or gender incongruence (ICD-11)
2. the pursuit of hormone therapy
3. native German speakers
4. age: 18-55
5. written informed consent following oral and written information
6. persons who are legally competent and mentally able to follow the instructions of the staff

Exclusion Criteria:

1. drug abuse/addiction
2. first-degree relatives with psychotic disorders
3. pregnant or breastfeeding
4. traumatic brain injuries
5. neurological diseases
6. known internal, e.g. metabolic, endocrine or cardiac disorders
7. magnetic metal implants
8. hearing disorders, voice disorders and pronounced hoarseness
9. shift workers or irregular day-night rhythm
10. persons placed in an institution by order of the authorities or courts
11. persons who are in a dependent or employment relationship with the auditor
12. simultaneous participation in a clinical trial
13. hormone treatment already started

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Transgender people seeking gender-affirming hormonal treatment who fullfill the inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-11-27 (Actual); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
changes in anatomical MRI | 7 minutes; assessed before gender affirming hormone therapy starts and 6 months after onset (corresponding time points are chosen for the healthy controls)
  measurment of anatomical differences between the groups and changes in the TG group throughout the gender-affirming hormone treatment
changes in Resting-state MRI measurements | 10 minutes; assessed before gender affirming hormone therapy starts and 6 months after onset
  measurment of resting-state activation differences between the groups and changes in the TG group throughout the gender-affirming hormone treatment
changes in Functional MRI measurements | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  measurment of activation differences during a voice and a face gender-recognition task between the groups and changes in the TG group throughout the gender-affirming hormone treatment
changes in self-ratings regarding quality of life throughout gender-affirming hormone treatment : WHOQoL-BREF | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  items regarding different aspects of daily life, 5-point likert scale, changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding quality of life throughout gender-affirming hormone treatment: Gender Congruence and Life Satisfaction Scale | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  items regarding influence of gender congruence on different aspects of daily life, 5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Brief Symptom Inventory | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  occurence of different symptoms during the last week, 5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
self-ratings regarding psychological well-being and psychiatric: Childhood Trauma Questionnaire | 1 hour; assessed before gender affirming hormone therapy starts
  5-point likert scale
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: ENRICHD Social Support Inventory | 1 hour; assessed before gender affirming hormone therapy starts and 1, 2, 4 and 6 months after onset
  5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Positive and negative affect scale | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Patient Health Questionnaire-9 | 1 hour; assessed before gender affirming hormone therapy starts and 1, 2, 4 and 6 months after onset
  items regarding depressive symptoms, 4-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding personality throughout gender-affirming hormone treatment: Personality Inventory for DSM-5 Brief Form | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  4-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Rosenberg Self-Esteem Scale | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  4-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Stait-Trait-Angst Inventar | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  4-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over timechanges are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Stress- and Coping Inventar | 1 hour; assessed before gender affirming hormone therapy starts and 1, 2, 4 and 6 months after onset
  7-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding psychological well-being and psychiatric Symptoms throughout gender-affirming hormone treatment: Strukturiertes Klinisches Interview für DSM 5 | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  interview conducted by investigator with questions regarding symptoms of different psychiatric disorders; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding sexuality throughout gender-affirming hormone treatment: Multidimensional Sexuality Questionnaires | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  items regarding sexual relationships, 5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding gender congruence throughout gender-affirming hormone treatment:Transgender Congruence Scale | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  5-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding sex roles throughout gender-affirming hormone treatment: Assessment of Gender-Related Attributes | 1 hour; assessed before gender affirming hormone therapy starts and 2, 4 and 6 months after onset
  items regarding typicale male and female personality traits, cognition and interests, 7-point likert scale
changes in self-ratings regarding sex roles throughout gender-affirming hormone treatment: Bem Sex Role Inventory | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  7-point likert scale; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in self-ratings regarding percpetion of and satisfaction with own body throughout gender-affirming hormone treatment : Fragebogen zur Beurteilung des eigenen Körpers | 1 hour; assessed before gender affirming hormone therapy starts and 6 months after onset
  each item has to be rated as false or true, resulting in scores for the dimensions self-esteem, insecurities and external appearance; changes are measured for TG, CG are used as a control for potential natural changes over time
changes in Hormone/protein analyses throughout gender-affirming hormone treatment | 5 minutes; assessed before gender affirming hormone therapy starts and 6 months after onset
  (free) testosterone, estradiol, progesterone, BDNF; changes are measured for TG, CG are used as a control for potential natural changes over time

CONTACTS AND LOCATIONS:
Overall Officials: Ute Habel, Prof. Dr., Study Director — Uniklinkum Aachen; Birgit Derntl, Prof. Dr., Study Director — Uniklinikum Tübingen
Locations (2):
- Germany (2):
  - Uniklinik RWTH Aachen, Aachen
  - Universitätsklinikum Tübingen, Tübingen

IPD SHARING:
Plan to Share IPD: Undecided